CLINICAL TRIAL: NCT04128254
Title: A Prospective Study in Chinese Patients With Lower Extremity Ankle Fracture of Oral Anticoagulants to Prevent Venous Thromboembolism (VTE)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-CPAFVTE
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Foot Ankle Injuries; Anticoagulants and Bleeding Disorders; Venous Thromboembolism
MeSH Terms: conditions — Hemostatic Disorders; Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental)
  Interventions: Drug: Apixaban Oral Tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Apixaban Oral Tablet

INTERVENTIONS:
Drug: Apixaban Oral Tablet — Apixaban is a kind of oral anticoagulant drugs used to prevent venous thromboembolism

SUMMARY:
Deep vein Thrombosis (Deep Venous Thrombosis, DVT) and Pulmonary Embolism, Pulmonary Embolism, PE) both collectively known as Venous thromboembolism (VTE) (Venous Thrombus Embolism, VTE), is a common clinical disease, and tremendous harmful. Ankle fractures in patients requiring long-term bed braking, increase the incidence of lower extremity deep vein thrombosis, anticoagulant therapy as an important measures to prevent thrombosis in clinical widely accepted, however, the literature anticoagulation effect incision healing. Whether to strike a balance between the two, to develop a foot fracture in accordance with the Chinese characteristics of anticoagulant solution is we try to solve the problem. The purpose of this study is aimed at the use of oral anticoagulants and physical anticoagulant treatment knee far foot fracture patients randomized controlled studies in China.

ELIGIBILITY:
Inclusion Criteria:

* (1) year full 18 one full year of life (2) one side of ankle fractures, calcaneal fractures, the metatarsal bone fracutures will use the internal fixation treatment 3) participants must be able to normal conversation, and understand the problems in the "subject subjective questionnaire", and could provide feedback using the appropriate language.

Exclusion Criteria:

* 1)Subjects did not provide a voluntary agreement 2) subjects participating in clinical research for pregnant or lactating women 3) has preoperative examination in the diagnosis of venous thromboembolism (VTE) 4) in patients with preoperative oral antiplatelet/anticoagulation drugs for a long time.

  5) surgery time fractures occur over time more than 3 weeks 6) patients exist pilon fractures (AO type 43-43 - B and C) and ankle multiple fractures, 7) pathological fractures (e.g., primary or metastatic tumors) 8) severe soft tissue injuries, open fractures or vascular injury or the combining bone fascia room syndrome; 9) multiple injuries, judge doesn't fit into the study by researchers, and other parts of the three or more than fracture 10) revision surgery (e.g., malunion, bone nonunion or infection) 11) merger of anticoagulant taboo disease, judge doesn't fit into the study by researchers, such as the active bleeding and clotting disorders, severe head trauma or acute spinal cord injury, platelet count < 20 ╳ 109 / L, etc.; 12) patients with anesthesia and surgery patients with contraindications to 13) on pp shaaban drug allergy 14) patients may be poor compliance, the researchers determined doesn't fit into the daily (such as excessive drinking or smoking, taking drugs) 15) patients in the past three months participated in other clinical trials; 16) in patients with poor compliance, judge not according to the study by the researchers plan to complete the test, such as schizophrenia and dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
the rate of venous thromboembolism (VTE) on 12th postoperative week | 12th postoperative week
  For individual subjects, if after 12 weeks to satisfy all of the following conditions, is considered an effective means to test: 1. The local infection, wound dehiscence, bleeding and swelling, local no abnormal activities; 2. Confirmed by doppler ultrasound has no lower limb venous thromboembolism (VTE); 3. No serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: SAHZJU, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No